CLINICAL TRIAL: NCT01123837
Title: A Closer Look at the Effect of Dextrose on Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Richard Applegate, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5100086
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D5LR (Active Comparator): In the treatment group, a 250cc bolus over 2 hrs of D5LR will be initiated prior to the end of surgery and continued in PACU.Blood glucose will be measured at 3 different timepoints using a point of care testing device (Accu-Chek). We will be measuring changes in blood glucose levels associated with PONV and the type and number of rescue medicines given at 30, 60, and 120 minutes after anesthesia and the first postoperative morning
  Interventions: Other: Intravenous fluid; Other: D5LR or lactated ringers
- lactated ringers (Active Comparator): In the control group, a 250cc bolus over 2 hrs of LR will be initiated prior to the end of surgery and continued in PACU. Blood glucose will be measured at 3 different timepoints using a point of care testing device (Accu-Chek). We will be measuring changes in blood glucose levels associated with PONV and the type and number of rescue medicines given at 30, 60, and 120 minutes after anesthesia and the first postoperative morning.
  Interventions: Other: Intravenous fluid; Other: D5LR or lactated ringers

INTERVENTIONS:
Other: Intravenous fluid — The treatment group will receive a 250cc bolus over 2 hrs of D5LR prior to the end of surgery and continued in the PACU. Blood glucose will be checked 3 different times using an Accu-chek monitor along with the type and number of rescue medications given at 30, 60, and 120 minutes after anesthesia and the post-op morning.
  The control group will receive a 250cc bolus over 2 hours of LR. Blood glucose will be monitored 3 times along with the type and how much of rescue medications are given at 30, 60 and 120 minutes post-op and the morning after surgery.
Other: D5LR or lactated ringers — The purpose of the study is to see if giving dextrose fluid in the veins (IV) decreases the risk of postoperative nausea and vomiting (PONV) in female urologic, gynecologic and breast outpatient surgery patients and at what blood sugar level.
  The reason for this study is that IV dextrose may decrease the incidence of PONV and the use of medications to treat PONV, while leading to sooner discharge after surgery. This can decrease overall healthcare cost and improving patient satisfaction.

SUMMARY:
"The purpose of this investigator-initiated study is to see if giving dextrose fluid in the veins (IV) decreases the risk of postoperative nausea and vomiting (PONV) in female urologic, gynecologic and breast outpatient surgery patients and at what blood surgery level. The reason for this study is that IV dextrose has been shown to decrease the incidence of PONV and the use of medications to treat PONV, while leading to sooner discharge after surgery. This can decrease overall healthcare cost and improving patient satisfaction."

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II
2. female urologic, gynecologic and breast surgery patients undergoing scheduled same day procedures at LLUMC Heart and Surgical Hospital

Exclusion Criteria:

1. age <18 or >65;
2. severe hypertension,diabetes mellitus, significant hepatic or renal disease
3. excessive blood loss
4. sustained (>10 min)>20% from baseline drop in BP after treatment
5. inability to follow protocol
6. refusal to sign consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
A Closer Look at the Effect of Glucose on Postoperative Nausea and Vomiting | approximately 24 hours
  The primary outcome measures will be the severity and incidence of PONV along with the type and number of rescue medications given at 0,30,60, and 120 minutes PACU time and the next morning.

SECONDARY OUTCOMES:
A Closer Look at the Effect of Dextrose on Post-operative nausea and vomiting | approximately 24 hours
  Secondary endpoints recorded will be length of surgery, history of PONV, amount of pain medicine administered, blood loss, drop in BP > 20%, unplanned hospital admission for PONV, and time till ready for discharge from PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Applegate, M.D., Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center Heart and Surgical Hospital, Loma Linda, California, United States